CLINICAL TRIAL: NCT03385564
Title: An Exploratory Maintenance Trial Evaluating the Effect of BI 655064 in Lupus Nephritis Patients Who Have Achieved a Meaningful Response Either at the End of 1293.10 or After an Induction Treatment Outside of 1293.10
Brief Title: An Exploratory Maintenance Trial of BI 655064 in Patients With Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1293-0013; 2017-003101-17 (EudraCT Number)
Record Dates: First submitted 2017-12-21; First posted 2017-12-28 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — BI 655064

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 655064 120 mg (Experimental): 120 milligrams (mg) BI 655064 were administered as solution for subcutaneous injection in a prefilled syringe once every 2 weeks plus the administration of matching placebo as subcutaneous injection in a prefilled syringe once every 2 weeks (in the alternative weeks without BI 655064 administration) over a treatment period of 52 weeks, followed by a 12-week follow-up period. The patients received 1 injection per week.
  Interventions: Drug: BI 655064
- Placebo (Placebo Comparator): Matching placebo were administered as solution for subcutaneous injection in a prefilled syringe once every week over a treatment period of 52 weeks, followed by a 12-week follow-up period. The patients received 1 injection per week.
  Interventions: Drug: Placebo
- BI 655064 180 mg (Experimental): 180 milligrams (mg) BI 655064 were administered as solution for subcutaneous injection in a prefilled syringe once every 2 weeks plus the administration of matching placebo as subcutaneous injection in a prefilled syringe once every 2 weeks (in the alternative weeks without BI 655064 administration) over a treatment period of 52 weeks, followed by a 12-week follow-up period. The patients received 1 injection per week.
  Interventions: Drug: BI 655064
- BI 655064 240 mg (Experimental): 120 milligrams (mg) BI 655064 were administered as solution for subcutaneous injection in a prefilled syringe once every week (240 mg every 2 weeks) over a treatment period of 52 weeks, followed by a 12-week follow-up period. The patients received 1 injection per week.
  Interventions: Drug: BI 655064

INTERVENTIONS:
Drug: BI 655064 — subcutaneous injection
  Arms: BI 655064 120 mg; BI 655064 180 mg; BI 655064 240 mg
Drug: Placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to evaluate the long term efficacy and safety of different doses of BI 655064 versus placebo as add-on therapy to Standard of Care (SOC) during maintenance therapy for lupus nephritis.

DETAILED DESCRIPTION:
Initially planned participating countries:

Argentina, Australia, Canada, Colombia, Czech Republic, France, Germany, Greece, Hong Kong, Italy, Japan, Republic of Korea, Malaysia, Mexico, Philippines, Poland, Portugal, Serbia, Spain, Taiwan, Thailand, United Kingdom, United States

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* Women of childbearing potential and men able to father a child must be ready and able to use two reliable methods of birth control simultaneously, one of which must be highly effective. Highly effective birth control per International Conference on Harmonisation (ICH) M3(R2) is a method that result in a low failure rate of less than 1% per year when used consistently and correctly. The reliable methods of birth control must be used before starting Mycophenolate mofetil/Azathioprine (MMF/AZA) and the trial drug; then continue during the trial period; and for at least 50 days after the last dose of MMF/AZA and trial medication. In case a female patient is treated with AZA the contraception shall continue for 90 days after treatment with AZA.A list of contraception methods meeting these criteria is provided in the patient information.
* Sexually active men must be ready to use condoms during treatment with MMF/AZA and for at least 90 days after cessation of MMF/AZA.
* Permanent sterilisation methods include hysterectomy, bilateral oophorectomy and bilateral salpingectomy.
* Tubal ligation is NOT a method of permanent sterilisation.
* A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

For Group 1 patients only:

- Achieved either a Complete renal Response (CRR) or a Partial Renal Response (PRR) or proteinuria ≤ 1g/d (or UP/UC ≤ 1) at the end of 1293.10.

Exclusion Criteria:

* Evidence of current or previous clinically significant diseases or medical conditions other than lupus, or findings of the medical examination (including vital signs and ECG) that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied.
* Significant central nervous system symptoms related to Systemic Lupus Erythematosus (SLE) based on investigators assessment.
* Clinically important acute or chronic infections including but not limited to HIV, hepatitis B or C.
* Impaired hepatic function defined as serum Aspartate Aminotransferase/Alanine Aminotransferase (AST/ALT), bilirubin or alkaline phosphatase > 2 x Upper Limit of Normal (ULN).
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 at screening (using CKD-EPI formula).
* Known hypersensitivity to any constituents of the trial medication; and/or contraindications to Mycophenolate mofetil (MMF) or Azathioprine (AZA) or glucocorticoids.
* The use of any restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Unable to comply with the protocol in the investigator's opinion.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (4):
  - Integral Rheumatology and Immunology Specialist, Plantation, Florida
  - Northwell Health, Great Neck, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
- Princess Alexandra Hospital, Woolloongabba, Australia
- CHU de Quebec-Universite Laval Research Centre, Québec, Canada
- Czechia (2):
  - General University Hospital, Prague
  - Institute of Rheumathology Prague, Prague
- Germany (2):
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
- Greece (2):
  - University General Hospital Attikon, Athens
  - University General Hospital of Heraklion, Heraklion, Crete
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Japan (4):
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
- Hospital Tengku Ampuan Rahimah, Klang, Malaysia
- Mexico (3):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Instituto Nacional de Cs Médicas y Nutrición S Zubiran, Mexico City
- Philippines (2):
  - Southern Philippines Medical Center, Davao City
  - Mary Mediatrix Medical Center, Lipa City, Batangas
- Poland (3):
  - University Clinical Hospital in Bialystok I, Bialystok
  - Norbert Barlicki University Clinical Hospital No.1, Lodz, Lodz
  - NZOZ Centrum Medyczne AESKULAP,Private Prac, Radom, Radom
- Portugal (2):
  - Hospital Curry Cabral, EPE, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
- Ajou University Hospital, Suwon, South Korea
- Thailand (4):
  - Siriraj Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Chiangmai University, Chiang Mai
  - Pramongkutklao Hospital, Rajathevee
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to evaluate long-term efficacy and safety of different doses of BI 655064 versus placebo as add-on therapy to standard of care during maintenance treatment for lupus nephritis.
Pre-assignment Details: This is an extension trial with the requirement to entry that subjects responded to treatment in 1293.10 (NCT02770170) and had the desire to continue participation in a clinical trial. Subjects were screened for eligibility prior to participation in trial 1293.10 (NCT02770170).
Period: Overall Study
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Started | 7 | 15 | 21 | 26
Intent to Treat Set | 7 | 15 | 21 | 26
Completed (Completed trial medication) | 7 | 14 | 16 | 17
Not Completed | 0 | 1 | 5 | 9
Not completed — Adverse Event | 0 | 0 | 3 | 3
Not completed — Other than listed | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): this patient set included all patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo | Total
Number analyzed (Participants) | 7 | 15 | 21 | 26 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.9 (6.5) | 36.5 (8.7) | 35.4 (10.5) | 34.8 (10.9) | 35.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 19 | 24 | 61
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 6 | 6 | 19
  Not Hispanic or Latino | 4 | 11 | 15 | 20 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 6 | 9 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 9 | 11 | 15 | 38
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Renal Response (CRR) and Without Any Renal Flares
Description: The adjusted (model-based, adjusted for race and proteinuria at screening) percentage of patients with complete renal response (CRR) and without any renal flares is reported. A logistic regression model was used including treatment and the covariates: race (Asian versus (vs.) non-Asian) and proteinuria <3 gram (g)/day vs. ≥3 g/day (or Urine protein (UP)/ Urine creatinine (UC) <3 vs. UP/UC ≥3) at screening.
  Complete renal response (CRR) was defined as urine protein (UP) < 0.5 g/day and either estimated glomerular filtration rate (eGFR) within normal range or decrease in eGFR < 20% from baseline if eGFR was below normal range (below lower limit of normal [LLN], where LLN = 90 mL/min.
Time Frame: At Week 52
Population: Intent to treat (ITT) set: this patient set included all patients from the treated set (TS) who had a baseline proteinuria (spot urine could be a used if the patient did not have 24 hours urine collections) and a baseline Estimated glomerular filtration rate (eGFR) value. Only subjects with non-missing results were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 20 | 25
Percentage of participants | 51.83 | 48.15 | 59.49 | 57.51
Statistical Analysis 1: Comparison: BI 655064 120 mg vs Placebo; Test type: Other — Percentage of patients with CRR at Week 52 without renal flare were analysed using a logistic regression model. Factors in the model included treatment and the covariates: race (Asian versus (vs.) non-Asian) and proteinuria <3 gram (g)/day vs. ≥3 g/day (or Urine protein (UP)/ Urine creatinine (UC) <3 vs. UP/UC ≥3) at screening; p = 0.7957, Regression, Logistic; Difference = -5.68, 80% CI 2-sided [-34.192 to 22.825] — The difference was calculated as value from BI 120 milligrams group minus value from Placebo group. Confidence intervals calculated using the delta method
Statistical Analysis 2: Comparison: BI 655064 180 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5811, Regression, Logistic; Difference = -9.37, 80% CI 2-sided [-31.178 to 12.440] — The difference was calculated as value from BI 180 milligrams group minus value from Placebo group. Confidence intervals calculated using the delta method
Statistical Analysis 3: Comparison: BI 655064 240 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8972, Regression, Logistic; Difference = 1.97, 80% CI 2-sided [-17.534 to 21.480] — The difference was calculated as value from BI 240 milligrams group minus value from Placebo group. Confidence intervals calculated using the delta method

2. Secondary Outcome: Percentage of Patients With Confirmed Complete Renal Response (CRR) and Without Any Renal Flares
Description: The percentage of patients with confirmed complete renal response (CRR) (defined as CRR at both Week 42 and Week 52 using urine protein (UP)/urine creatine (UC) ratio [UP/UC] from the spot urines) and without any renal flares is reported. Complete renal response (CRR) was defined as urine protein (UP) < 0.5 g/day and either estimated glomerular filtration rate (eGFR) within normal range or decrease in eGFR < 20% from baseline if eGFR was below normal range (below lower limit of normal [LLN], where LLN = 90 mL/min).
Time Frame: At Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 13 | 20 | 25
Percentage of participants | 42.9 | 30.8 | 50.0 | 52.0
Statistical Analysis 1: Comparison: BI 655064 120 mg vs Placebo; Test type: Other; p = 0.8250, Barnard test; Difference = -9.14, 80% CI 2-sided [-32.83 to 17.02] — The difference was calculated as value from BI 120 milligrams group minus value from Placebo group. Confidence intervals calculated using the Newcombe method
Statistical Analysis 2: Comparison: BI 655064 180 mg vs Placebo; Test type: Other; p = 0.2562, Barnard test; Difference = -21.23, 80% CI 2-sided [-39.44 to 0.51] — The difference was calculated as value from BI 180 milligrams group minus value from Placebo group. Confidence intervals calculated using the Newcombe method
Statistical Analysis 3: Comparison: BI 655064 240 mg vs Placebo; Test type: Other; p = 0.9632, Barnard test; Difference = -2.00, 80% CI 2-sided [-20.45 to 16.62] — The difference was calculated as value from BI 240 milligrams group minus value from Placebo group. Confidence intervals calculated using the Newcombe method

3. Secondary Outcome: Percentage of Patients With Proteinuria <0.8 Grams (g)/Day (d) and Without Any Renal Flares at Week 52
Description: The percentage of patients with proteinuria <0.8 grams (g)/day (d) and without any renal flares at week 52 is reported.
Time Frame: At Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 20 | 25
Percentage of participants | 57.1 | 50.0 | 60.0 | 60.0
Statistical Analysis 1: Comparison: BI 655064 120 mg vs Placebo; Test type: Other; p = 0.9275, Barnard test; Difference = -2.86, 80% CI 2-sided [-28.58 to 21.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 655064 180 mg vs Placebo; Test type: Other; p = 0.6064, Barnard test; Difference = -10.00, 80% CI 2-sided [-29.90 to 10.64] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: BI 655064 240 mg vs Placebo; Test type: Other; Difference = 0.00, 80% CI 2-sided [-18.37 to 18.07] — [estimate comment as in outcome 2, analysis 3]

4. Secondary Outcome: Percentage of Patients With Complete Renal Response (CRR) at Week 52 and Sustained Steroid Reduction to ≤5 Milligrams (mg)/Day (d) From Week 26 to Week 52
Description: The percentage of patients with complete renal response (CRR) at Week 52 and sustained steroid reduction to ≤5 milligrams (mg)/day (d) from Week 26 to Week 52 is reported. Complete renal response (CRR) was defined as urine protein (UP) < 0.5 g/day and either estimated glomerular filtration rate (eGFR) within normal range or decrease in eGFR < 20% from baseline if eGFR was below normal range (below lower limit of normal [LLN], where LLN = 90 mL/min.
Time Frame: At Week 52 (Sustained Steroid Reduction to ≤5 mg/d was evaluated from Week 26 to Week 52).
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 18 | 23
Percentage of participants | 42.9 | 42.9 | 55.6 | 39.1
Statistical Analysis 1: Comparison: BI 655064 120 mg vs Placebo; Test type: Other; p = 0.9119, Barnard test; Difference = 3.73, 80% CI 2-sided [-20.53 to 29.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 655064 180 mg vs Placebo; Test type: Other; p = 0.8510, Barnard test; Difference = 3.73, 80% CI 2-sided [-16.58 to 24.31] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: BI 655064 240 mg vs Placebo; Test type: Other; p = 0.3498, Barnard test; Difference = 16.43, 80% CI 2-sided [-3.53 to 34.73] — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Percentage of Patients Experiencing at Least One Renal Flare During 52 Weeks
Description: The percentage of patients experiencing at least one renal flare during 52 weeks is reported.
Time Frame: At Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 21 | 25
Percentage of participants | 0 | 21.4 | 0 | 16.0
Statistical Analysis 1: Comparison: BI 655064 180 mg vs Placebo; Test type: Other; p = 0.7921, Barnard test; Difference = 5.43, 80% CI 2-sided [-10.19 to 23.57] — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Time to First Renal Flare Over the Course of 52 Weeks
Description: The time to first renal flare over the course of 52 weeks is reported.
Time Frame: Up to 52 weeks.
Population: Intent to treat (ITT) set: this patient set included all patients from the treated set (TS) who had a baseline proteinuria (spot urine could be a used if the patient did not have 24 hours urine collections) and a baseline Estimated glomerular filtration rate (eGFR) value. Only subject with non-missing results were included in the analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 4
Weeks |  | 36.0 [26 to 52] |  | 37.5 [6 to 52]

7. Secondary Outcome: Percentage of Patients With Partial Renal Response (PRR) and Without Any Renal Flares Derived From Urine Protein (UP) 24 Hours (h) Collection at Week 52
Description: The percentage of patients with partial renal response (PRR) and without any renal flares derived from urine protein (UP) 24 hours (h) collection at Week 52 is reported. Partial renal response (PRR) was defined as at least 50% reduction of proteinuria from baseline if estimated glomerular filtration rate (eGFR) was within normal range at time of assessment or decrease of eGFR <20% from baseline if eGFR was below normal range at time of assessment.
Time Frame: At Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 20 | 25
Percentage of participants | 100.0 | 64.3 | 75.0 | 68.0
Statistical Analysis 1: Comparison: BI 655064 120 mg vs Placebo; Test type: Other; p = 0.1016, Barnard test; Difference = 32.00, 80% CI 2-sided [10.28 to 44.74] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 655064 180 mg vs Placebo; Test type: Other; p = 0.8323, Barnard test; Difference = -3.71, 80% CI 2-sided [-23.79 to 15.29] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: BI 655064 240 mg vs Placebo; Test type: Other; p = 0.6247, Barnard test; Difference = 7.00, 80% CI 2-sided [-10.50 to 23.31] — [estimate comment as in outcome 2, analysis 3]

8. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Total Score at Week 12
Description: Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score at Week 12 is reported. Change from baseline at Week 12 is calculated as: value at Week 12 - value at baseline. SLEDAI assessment consists of 24 items capturing non-renal and renal symptoms. The total score captures non-renal and renal symptoms. Each of the 24 items has a score ranging from 1 to 8. A participant will get the score if the event of the item presents, while 0 if not. 8 items have the score 8, 6 items have the score 4, 7 items have the score 2, and 3 items have the score 1. The SLEDAI Total score is the sum of the scores of the 24 items, ranging from 0 (better health) to 105 (worse health).
Time Frame: At baseline and at Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 13 | 18 | 25
Score on a scale | -8.4 (5.8) | -7.5 (4.3) | -9.3 (4.9) | -7.7 (6.1)

9. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Total Score at Week 26
Description: Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score at Week 26 is reported. Change from baseline at Week 26 is calculated as: value at Week 26 - value at baseline. SLEDAI assessment consists of 24 items capturing non-renal and renal symptoms. The total score captures non-renal and renal symptoms. Each of the 24 items has a score ranging from 1 to 8. A participant will get the score if the event of the item presents, while 0 if not. 8 items have the score 8, 6 items have the score 4, 7 items have the score 2, and 3 items have the score 1. The SLEDAI Total score is the sum of the scores of the 24 items, ranging from 0 (better health) to 105 (worse health).
Time Frame: At baseline and at Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 16 | 21
Score on a scale | -8.7 (5.7) | -7.9 (3.5) | -11.3 (4.8) | -5.9 (5.2)

10. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Total Score at Week 42
Description: Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score at Week 42 is reported. Change from baseline at Week 42 is calculated as: value at Week 42 - value at baseline. SLEDAI assessment consists of 24 items capturing non-renal and renal symptoms. The total score captures non-renal and renal symptoms. Each of the 24 items has a score ranging from 1 to 8. A participant will get the score if the event of the item presents, while 0 if not. 8 items have the score 8, 6 items have the score 4, 7 items have the score 2, and 3 items have the score 1. The SLEDAI Total score is the sum of the scores of the 24 items, ranging from 0 (better health) to 105 (worse health).
Time Frame: At baseline and at Week 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 5 | 7 | 9 | 13
Score on a scale | -6.6 (3.4) | -6.3 (2.4) | -11.1 (5.1) | -6.5 (6.7)

11. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Total Score at Week 52
Description: Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score at Week 52 is reported. Change from baseline at Week 52 is calculated as: value at Week 52 - value at baseline. SLEDAI assessment consists of 24 items capturing non-renal and renal symptoms. The total score captures non-renal and renal symptoms. Each of the 24 items has a score ranging from 1 to 8. A participant will get the score if the event of the item presents, while 0 if not. 8 items have the score 8, 6 items have the score 4, 7 items have the score 2, and 3 items have the score 1. The SLEDAI Total score is the sum of the scores of the 24 items, ranging from 0 (better health) to 105 (worse health).
Time Frame: At baseline and at Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
Number analyzed (Participants) | 7 | 14 | 16 | 17
Score on a scale | -8.9 (6.1) | -7.2 (4.0) | -10.6 (4.9) | -5.3 (8.0)

ADVERSE EVENTS:
Time Frame: For serious and non-serious adverse events: From first dose of trial medication until last dose + 50 days of residual effect period, up to 52 weeks + 50 days. For all-cause mortality: From first dose of trial medication until end of study, up to 64 weeks.
Description: Treated set (TS): this patient set included all patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Arm/Group | BI 655064 120 mg | BI 655064 180 mg | BI 655064 240 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/15 | 1/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/15 | 6/21 | 4/26
Other Adverse Events (participants affected / at risk) | 6/7 | 11/15 | 15/21 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655064 120 mg (N=7) | BI 655064 180 mg (N=15) | BI 655064 240 mg (N=21) | Placebo (N=26)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis of central nervous system (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ocular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655064 120 mg (N=7) | BI 655064 180 mg (N=15) | BI 655064 240 mg (N=21) | Placebo (N=26)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0
Visual field defect (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 5 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Blood lactate dehydrogenase decreased (Investigations) | 1 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 2 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 3
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT03385564/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03385564/SAP_001.pdf